CLINICAL TRIAL: NCT03795077
Title: Effect of a Higher Education Programme Based on Professional Ethics in Physiotherapy Students
Brief Title: Effect of a Programme Based on Professional Ethics in Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, PhD, PT, assisstant professor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 545879652
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Ethics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group followed traditional lectures about professional ethics during 3 months as usual.
- Experimental group (Experimental): Experimental group followed the programme based in professional ethics. A specific syllabus about Professional Ethics was developed. It consisted of 6 themes and included topics as moral values, ethics and moral, bioethics and professional ethics, ecc. Six related activities were created: to solve situations related to real clinical practices. Face to face group sessions based on cooperative learning were planned. Students were divided in small groups, and active participation techniques were used. Techniques used: concept maps, glossaries, brainstorming, four corners activity, aquarium, philip 6-6, kahoot, Realm Individual-Process Situation, reduced groups, guided debates, and discussion groups.
  Interventions: Other: Experimental group

INTERVENTIONS:
Other: Experimental group — Experimental group followed the 3-months programme based in professional ethics. A specific syllabus about Professional Ethics was developed. It consisted of 6 themes and included topics as moral values, ethics and moral, bioethics and professional ethics, ecc. Six related activities were created: to solve situations related to real clinical practices. Face to face group sessions based on cooperative learning were planned. Students were divided in small groups, and active participation techniques were used.
  Arms: Experimental group

SUMMARY:
The aim of this study was to assess the effect of a higher education programme based on professional ethics in physiotherapy students.

A simple-blind clinical trial was performed. A three-months program based in professional ethics was carried out.

The investigators compared a control group (traditonal lectures) with an intervention group (syllabus, activities, face to face techniques). Students´ attitudes, knowledge, professional values, and opinions towards professional ethics were evaluated before and after the programme, in both groups. All participants were informed about the study and procedures, and provided written informed consent.

DETAILED DESCRIPTION:
Participants. Second-year degree students of Physiotherapy Degree at the University, aged between 20 and 30 years, were recruited voluntarily from January 2019 to April 2019 . All enrolled participants were informed of the purpose of the study and procedures, and provided written informed consent. The study was carried out at the institution where the authors belong.

Research design. A prospective simple-blind trial was performed. After baseline assessment, participants were allocated to one of the two groups (control group and experimental group). An external assistant not involved in the study performed assignment.

Intervention. A Physiotherapy professor with over-10-year experience in Ethics and Physiotherapy performed the teaching methodology and opened the allocation envelopes and applied the teaching methodology to the EG according to the group assignment. The intervention consisted of a three-month program based in professional ethics, including two phases: A) syllabus and activities; and B) face to face group sessions including techniques such as concept maps, glossaries, brainstorming, four corners activity, aquarium, philip 6-6, kahoot, Realm Individual-Process Situation, reduced groups, guided debates, and discussion groups.

ELIGIBILITY:
Inclusion Criteria:

* To study the physical therapy degree at the University of Valencia

Exclusion Criteria:

* Exclusion criterion was having prior training on Ethics subject

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Knowledge of Professional Ethicss | 12 weeks
  measured with an ad-hoc retention test. The students were not previously informed about retention exams to avoid any preparation for the test. The tests included 15 multiple choice questions that assessed basic professional ethics concepts that physiotherapy students are required to know, such as: moral values, bioethics and Professional Ethics in physiotherapy, professional ethical principles, physiotherapists deontological code, ethical situations, or professional values in physiotherapy.

SECONDARY OUTCOMES:
Perception of knowledge regarding professional Ethics | 12 weeks
  A self-reported questionnaire of 19 items (the Perceptions about Knowledge regarding Professional Ethics in Physiotherapy, PKPEPT, Cronbach's alpha=0.760) was previously described.27,28 The higher score indicated the best perception of knowlegde. The questionnaires' items included basic professional ethics concepts that physiotherapy students are required to know. Therefore, questions assessed participants' perception about knowledge regarding basic concepts in Professional Ethics and their application in physiotherapy care. Items were created in order to be important and to be clearly related with perception of knowledge.
Quality assessment | 12 weeks
  It was assessed for both groups by the Teaching evaluation of the Center for Quality of the University of Valencia. This center offers the students online surveys with different items evaluating the teaching methodologies, materials and general satisfaction by a Likert scale (1 totally disagree to 5 totally agree) in undergraduate degree, through the Virtual Office of the University.
Satisfaction assessment | 12 weeks
  For the Cooperative Learning group, an ad-hoc satisfaction questionnaire was carried out, using the Kahoot application. The satisfaction questionnaire included 16 questions in total: 5 dichotomous questions about opinion about the methodology, 5 dichotomous questions about the themes; 3 Likert-type questions (not at all / little / quite / a lot) about interest and usefulness of the content / contents, and 3 questions about satisfaction, usefulness and fun with respect to the techniques used, Likert-type: from 0 to 5 points. This evaluation was only carried out at the end of the program.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No